CLINICAL TRIAL: NCT05415657
Title: Denosumab Protects Bone Loss and Function in Osteopenia Patients With Lumbar Degenerative Diseases After Lumbar Fusion Surgery, a Randomized, Placebo Controlled Trial.
Brief Title: Denosumab Effect on Bone Quality and Function After Lumbar Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ShenzhenPH spine01
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Osteopenia; Spine Fusion; Denosumab Allergy
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Denosumab; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): Denosumab 60 mg were injected subcutaneously Q6M on the same day after lumbar fusion surgery, and all patients received calcium supplementation 1200 mg/D and vitamin D 800 IU/D.
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Equal volume of saline (0.9%) as placebo were injected subcutaneously Q6M on the same day after lumbar fusion surgery, and all patients received calcium supplementation 1200 mg/D and vitamin D 800 IU/D.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab — Denosumab 60 mg per 6 month were injected subcutaneously on the same day after lumbar fusion surgery, and all participants received calcium supplementation 1200 mg/D and vitamin D 800 IU/D.
  Other Names: Denosumab 6 month/subcutaneous
  Arms: Denosumab
Drug: Placebo — Equal volume of saline (0.9%) as placebo Q6M were injected subcutaneously on the same day after lumbar fusion surgery, and all participants received calcium supplementation 1200 mg/D and vitamin D 800 IU/D.
  Other Names: Placebo 6 month/subcutaneous
  Arms: Placebo

SUMMARY:
Degenerative lumbar spinal diseases have become a common health problem and the most frequent indication for spinal surgery in elderly individuals. It mainly contain lumbar spinal stenosis and spondylolisthesis, occurs in most people over 60 years of age, and patients primarily diagnosed with lumbar degenerative disease are more likely to have osteoporosis. Our study was to explore denosumab effect on bone quality and functional status in osteopenia patients with lumbar degenerative diseases after lumbar fusion surgery.

DETAILED DESCRIPTION:
However, It was still unknown for denosumab effect on osteopenia patients after lumbar fusion. Bone mineral density(BMD), bone turnover marker, lumbar functional status Roland-Morris Disability Functioning Questionnaire (RMDQ) and quality of life EuroQol Five-Dimension (EQ-5D), and Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31) score, rate of new fracture, re-operation, lumbar fusion, complications or adverse events were still unknown. Our study will explore the effect of denosumab on lumbar, total hip, femoral neck BMD and bone turnover markers, functional status EQ-5D, QUALEFFO-31 and RMDQ score of participants after lumbar fusion at 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 40 to 85 years
* who diagnosed with lumbar spinal stenosis or lumbar spondylolisthesis
* osteopenia with BMD T score between -1.0 and -2.5 via dual-energy X-ray
* low back pain or leg numbness or weakness
* MRI demonstrated signs of nerve compression

Exclusion Criteria:

* cauda equina syndrome
* progressive neurologic deficit
* history of cancer
* scoliosis greater than 15°
* back open surgery history
* have contraindications for surgery
* who had anti-osteoporosis medication within 6 weeks

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Lumbar bone mineral density (BMD) | up to 12 months
  Lumbar vertebral (L1 to L4, except the surgery segment) BMD were determined at baseline, 6 and 12 months via Dual-energy X-ray.
Total hip BMD | up to 12 months
  Total hip BMD were determined at baseline, 6 and 12 months via Dual-energy X-ray.
Femoral neck BMD | up to 12 months
  Femoral neck BMD were determined at baseline, 6 and 12 months via Dual-energy X-ray.
Type 1 n-terminal propeptide P1NP | up to 12 months
  Bone formation marker, type 1 n-terminal propeptide P1NP were determined at baseline, 6 and 12 months after surgery.
C-terminal crosslinking type 1 collagen terminal peptide CTX | up to 12 months
  Bone resorption marker, C-terminal crosslinked type 1 collagen terminal peptide, CTX were assessed at baseline, 6 and 12 months after surgery.
Visual analog scale (VAS) back | up to 12 months
  VAS score for back pain were assessed at baseline, 6 and 12 months. Use a ruler about 10cm long, one side is marked with "0" and the other "10" respectively. A score of 0 indicates no pain, 10 indicates the most unbearable pain.
VAS leg | up to 12 months
  VAS score for leg pain were assessed at baseline, 6 and 12 months. Use a ruler about 10cm long, one side is marked with "0" and the other "10" respectively. A score of 0 indicates no pain, 10 indicates the most unbearable pain

SECONDARY OUTCOMES:
EQ-5D quality of life questionnaire | up to 12 month
  EQ-5D descriptive system is a preference-based quality of life measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. From this, a quality of life score can be calculated ranging from -0.594, indicating a health state worse than death where 0 is death, to 1, indicating full health
Roland-Morris Disability Questionnaire | up to 12 month
  The Roland-Morris Disability Questionnaire is a health status measure designed to be completed by patients to assess physical disability due to low back pain. The lowest score is 0, the highest 24. The higher the score, the more severe the dysfunction.
QUALEFFO-31 Questionnaire | up to 12 month
  QUALEFFO-31, which contains three domains including pain, physical function, and mental function. The worse the health related quality of life condition, the higher the score. This scale is assessed on a scale of 0 to 100, with 0 indicating the highest QoL and 100 the lowest.
Lumbar Fusion rate | up to 12 month
  We determined lumbar fusion rate via CT at 12 month after surgery.The lowest rate is 0, the highest 100%. The higher the score represents higher fusion rate.
New fracture rate | up to 12 month
  New fracture rate including new vertebral fracture and non-vertebral fracture was assessed at 12 month after surgery. The lowest score was 0, the highest score was 100%. The lower score represents no fracture.
Reoperation rate | up to 12 month
  Reoperation rate was assessed at 12 month after surgery. The lowest reoperation rate was 0, the highest score was 100%.
Complications | up to 12 month
  Complications such as cage subsidence, pedicle screw loosening, infection, peripheral nerve injury, recurrent symptoms were assessed at 12 months follow-up.
Adverse effect | up to 12 month
  The main adverse effect including deep vein thrombosis, rash, joint pain, headache, nausea, pneumonia, necrosis of jaw, atypical femoral fracture, pulmonary embolism, transfer to intensive care unit (ICU), stroke, acute renal failure, myocardial infarction and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- ShenzhenPH, Shenzhen, Guangdong, China